CLINICAL TRIAL: NCT06471400
Title: Developing Strategies to Facilitate Consent of Legally Authorized Representatives to Clinical Trials - a Prospective, Single-arm, Open-label Exploratory Trial
Brief Title: Developing Strategies to Facilitate Consent of Legally Authorized Representatives to Clinical Trials
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, PD Dr. Alexander Supady, Attending Physician, University Hospital Freiburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-1162-S1
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Critical Illness; Loss of Consciousness
MeSH Terms: conditions — Critical Illness; Unconsciousness | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient relative/LAR interview (Other): Study intervention: interview with patient relative/LAR
  Interventions: Other: interview

INTERVENTIONS:
Other: interview — patient relatives or legal authorized representatives will be interviewed

SUMMARY:
This study aims to gather insights into the perceptions of legal representatives regarding the recruitment process for clinical trials in the intensive care setting when the patients cannot decide for themselves. With this information, effective strategies will be developed to increase involvement and the feeling of ownership of LARs of (potential) participants in clinical trials and thus enhance and facilitate patient recruitment for clinical trials. The single-arm study design does not include a choice of comparator, as the focus of this trial is to explore the perceptions of the participants at first hand without comparing different cohorts or strategies.

DETAILED DESCRIPTION:
The evidence for specific therapies and treatment strategies, particularly for critically ill patients, remains limited. A significant difficulty for the planning, initiation and implementation of clinical trials in these patients is the urgency of the necessary medical measures, which leaves patients and their relatives, as well as the treating clinicians, little time and opportunities to present necessary studies and to inform the patients or their legal guardians about them. Critically ill patients are a particularly vulnerable group of patients. The measures required as part of a study can mean additional efforts for these patients over and above the burden of the disease and the necessary diagnostic and therapeutic measures, which are only justified if special duties of care are observed. In addition to an ethical assessment of the study, this also includes providing comprehensive information to patients or their legal representatives.

In this study, the process of informing and educating patients or their legal representatives will be examined in more detail. The aim of the study is to gain a better understanding of this process, in particular the perceptions and views of the persons to be informed, and specifically to investigate which aspects are particularly important to patients and their legal representatives in an information and education discussion and what information they need in order to be able to consider participating in a study or what reasons exist that would prevent them from giving their consent. The overall aim of this study is to improve the information and education process.

For some years now, the involvement of patients and relatives in individual aspects of the planning and conduct of clinical trials has been increasingly demanded and promoted. For example, large public funders often require the involvement of patient and/or family representatives at an early stage in the planning of trials. The objectives of this study are based on these expectations.

ELIGIBILITY:
Inclusion Criteria:

* The study will include LARs of adult patients aged 18 years or older who are admitted to the Freiburg University Medical Center in Germany.

Exclusion Criteria:

* LARs who have expressed their unwillingness to participate in the study or have objected to the measures implemented in the study will not be included.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-06-17 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
relative/LAR perception | actual day
  The primary aim of the study is to evaluate the perceptions of LARs towards the recruitment process for clinical trials. This is an exploratory examination. All findings are considered merely hypothesis generating and will be used for designing further trials based on sound hypotheses following the findings from this trial.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Supady, MD, Principal Investigator — Freiburg University Medical Center
Locations (1):
- Freiburg University Medical Center, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No